CLINICAL TRIAL: NCT00560339
Title: Does Lung Impedance Correlate With Changes in BNP in Stable and Acutely Decompensated Heart Failure Patients?
Acronym: IMPEDE-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southern New Jersey Cardiac Specialists (Other)
Collaborators: Medtronic (Industry)
Other Study IDs: 20051601
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-11

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Implantable Defibrillators; Intrathoracic Impedance
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether there is a relationship between serial B-natriuretic peptide (BNP) and implantable device measured intrathoracic impedance in symptomatic and asymptomatic heart failure patients over a 1-year period. Furthermore, this study will establish whether implantable device measured intrathoracic impedance trends with the distance walked on a six-minute hall walk (6MHW), an exercise-based acute measure that has also been associated with heart failure clinical status.

DETAILED DESCRIPTION:
This is a prospective non-randomized longitudinal study. One hundred subjects will participate in 6 monthly and 3 bi-monthly serial assessments of plasma-based BNP, implantable device measured intrathoracic impedance, and clinical evaluation of heart failure status. Each patient will be enrolled in the study for a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Baseline BNP > 80 pg/ml
* Meets current guidelines for ICD implantation with or without CRT
* Receiving a Medtronic InSync Sentry, Concerto, Virtuoso, or subsequently approved Medtronic ICD with the OptiVol feature.
* Walk < 450 meters during 6 minute hall walk test

Exclusion Criteria:

* Less than 18 years of age
* Life expectancy < 6 months
* History of non-compliance with clinic visits or study-related tasks which may decrease chance of completing of the study
* Physical disability which limits exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving with an implantable cardioverter defibrillator (ICD) with or without cardiac resynchronization therapy (CRT).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2005-09; Study Completion 2009-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Andriulli, DO, Principal Investigator — Southern New Jersey Cardiac Specialists
Locations (6):
- United States (6):
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Southern New Jersey Cardiac Specialists, Voorhees Township, New Jersey
  - St. Francis Hospital, Roslyn, New York
  - Carolinas Healthcare System/The Sanger Clinic, Charlotte, North Carolina
  - Mid State Cardiology Associates, Nashville, Tennessee
  - Medical College of Wisconsin /Froedtert Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Behnes M, Schmidberger M, Mashayekhi K, Vadala G, Moroni A, Guiterrez-Chico JL, Ayoub M, Christiansen EH, Pyxaras S, Bufe A, Krotz F, Schmitt A, Lau F, Reinhardt M, Forner J, Dudda J, Abel N, Hoepfner MK, Aubel C, Abumayyaleh M, Weidner K, Akin I, Schupp T. Coronary Chronic Total Occlusions Affect Long-Term Prognosis in Heart Failure With Mildly Reduced Ejection Fraction. J Am Heart Assoc. 2025 Sep 2;14(17):e042368. doi: 10.1161/JAHA.125.042368. Epub 2025 Aug 22. PMID 40847486